CLINICAL TRIAL: NCT00675896
Title: A Double Blind, Randomized Placebo Controlled Study of the Efficacy, Safety and Tolerability of Quetiapine Fumarate Sustained Release(Seroquel SRTM) in the Treatment of Major Depression With Comorbid Fibromyalgia Syndrome.
Brief Title: A Study of Quetiapine Fumarate Sustained Release in Major Depression With Comorbid Fibromyalgia Syndrome
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Dr Alexander McIntyre Inc. (Other)
Responsible Party: Dr Alexander McIntyre ., Dr Alexander McIntyre Inc.
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: D1443C00007; D1443C00007
Record Dates: First submitted 2008-05-08; First posted 2008-05-12 (Estimated); Last update posted 2011-07-06 (Estimated); Status verified 2011-07

CONDITIONS: Major Depression
Keywords: major depression with comorbid fibromyalgia.
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Quetiapine Fumarate Sustained Release(Seroquel SR)50 mg/day for the first 2 days and then up to 150mg/day. After two weeks the dose will be doubled up to 300mg at night at the discretion of the investigator, using patient tolerance and response as guidelines over the duration of the trial.
  Interventions: Drug: Quetiapine Fumarate Sustained Release
- 2 (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Quetiapine Fumarate Sustained Release — 50 mg/day for the first 2 days and then up to 150mg/day. After two weeks the dose will be doubled up to 300mg at night at the discretion of the investigator
  Other Names: Seroquel XR
  Arms: 1
Drug: Placebo — 1 tablet at HS for 2 days then 3 tablets at HS for 2 weeks
  Arms: 2

SUMMARY:
To compare the efficacy of Quetiapine SR versus placebo over 8 weeks in unipolar non-psychotic adult outpatients depression and comorbid fibromyalgia. This will be measured by the last observation carried forward (LOCF) mean change from baseline to week 8 on the Hamilton Depression Scale (HAM-D) total score.

For the purposes of this study, response regarding improvement in depressive symptoms will be defined as a 50% decrease in HAM-D scores over 8 weeks. Furthermore, proportion of patients achieving remission is defined as an HAM-D total score of 7 at end of treatment. The anxiety comorbid symptoms often associated with major depression will be assessed with the HAM-A (14 items) scale. Proportion of patients responding and achieving remission of anxiety symptoms are defined respectively as a reduction of 50% in the HAM-A total score from baseline and a HAM-A total score of 7 at the end of treatment.

DETAILED DESCRIPTION:
Secondary Endpoints include

* Change from baseline to week 8 in Brief Pain Inventory (short form) total score.
* Changes from baseline to week 8 in HAM-A total scores Changes from baseline to week 8 in CGI Severity of illness scores. Clinical Global Impression - Improvement (CGI-I) score from randomisation to Week 8 Change from baseline in the Fibromyalgia Impact Questionnaire (FIQ). Change from baseline in the Sleep Scale from the Medical Outcome Study (MOS). Change from baseline in the Sheehan Disability Scale (SDS). Change from baseline in the Quality of Life Enjoyment and Satisfaction Questionnaire- Short Form (Q-LES-Q-SF).

Change from baseline in the Patient Health Questionaire-15 (PHQ-15). Change from baseline in the Global Assessment Scale (GAS).

The side effects and the tolerability profiles of Quetiapine SR at the dose range used in the study will be assessed at every visit following the initial visit.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a DSM IV diagnosis of major depression and fibromyalgia confirmed by using the American College of Rheumatology criteria. Male or female between the ages of 18 and 65.
* Patients who score at least 22 on the 17-item HAM-D scale and at least 4 (i.e., moderately ill) on the Clinical Global Impression (CGI) severity scale. Both criteria have to be met at screening and baseline (Study Day 0).

Exclusion Criteria:

* Patients with DSM-IV Axis 1 disorder other than MDD and Chronic Pain Disorder within 6 months of enrolment.
* History of inadequate response to adequate treatment (6 weeks) with 2 or more classes of antidepressants during current depressive episode.
* Patients who, in the investigator's opinion, pose a risk for suicide.
* History of suicide attempt within 3 years of entering study.
* Current depressive episode secondary to general medical condition excluding Fibromyalgia.
* History or presence of bipolar disorder or psychosis.
* Post traumatic stress disorder, anorexia nervosa or bulimia nervosa.
* Patients with diagnosis of DSM-IV Axis II disorder which has a major impact on the patient's current psychiatric status.
* Present DSM IV diagnosis of substance abuse or dependence within 6 months prior of the screening visit (except dependence in full remission, and except caffeine, nicotine or opiate dependence)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2007-04; Primary Completion 2011-06 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
last observation carried forward (LOCF) mean change from baseline to week 8 on the Hamilton Depression Scale (HAM-D) total score. | 8 weeks

SECONDARY OUTCOMES:
Change from baseline to week 8 in: Brief Pain Inventory,HAM-A,CGI-S,FIQ, Sleep Scale from the Medical Outcome Study,SDS,QLES- Short Form,PHQ-15,Global Assessment Scale,Improvement (CGI-I) score from randomisation to Week 8 | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Alexander W McIntyre, FRCPC, Principal Investigator — Dr. A McIntyre Inc; Penticton Regional Hospital
Locations (1):
- Dr. A McIntyre Inc, Penticton, British Columbia, Canada

REFERENCES:
- [Derived] McIntyre A, Paisley D, Kouassi E, Gendron A. Quetiapine fumarate extended-release for the treatment of major depression with comorbid fibromyalgia syndrome: a double-blind, randomized, placebo-controlled study. Arthritis Rheumatol. 2014 Feb;66(2):451-61. doi: 10.1002/art.38228. PMID 24504819